CLINICAL TRIAL: NCT02909621
Title: Evaluation of Efficacy, Tolerance, and Dose Effects of a Curcuma Extract (FLEXOFYTOL®) Versus PLACEBO in Patients With Knee osteoARthritis (COPRA)
Brief Title: Evaluation of FLEXOFYTOL® Versus PLACEBO
Acronym: COPRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilman S.A. (Industry)
Collaborators: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: COPRA
Record Dates: First submitted 2016-09-13; First posted 2016-09-21 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis
Keywords: OsteoArthritis; FLEXOFYTOL®; Curcuma; biomarkers
MeSH Terms: conditions — Osteoarthritis | interventions — turmeric extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): Group A: FLEXOFYTOL® high dosage
  Interventions: Dietary Supplement: FLEXOFYTOL®
- Group B (Active Comparator): Group B: FLEXOFYTOL® low dosage
  Interventions: Dietary Supplement: FLEXOFYTOL®
- Group C (Placebo Comparator): Group C: PLACEBO
  Interventions: Other: PLACEBO

INTERVENTIONS:
Dietary Supplement: FLEXOFYTOL® — The product FLEXOFYTOL® is bio-optimized curcumin.
  Other Names: curcuma extract
  Arms: Group A; Group B
Other: PLACEBO
  Arms: Group C

SUMMARY:
This study is a prospective, randomized, double-blind, placebo-controlled with 3 parallel-groups and multicenter trial in patients suffering from knee OA (osteoarthrosis).

A first exploratory non comparative study (TILFLEXY002, NCT01909037, Henrotin et al., 2014 BMC Complementary and Alternative Medicine) evaluated the efficacy of FLEXOFYTOL® at the dose of 2x3 caps/day, during a 3-month period, in 22 patients suffering from knee OA, on the serum levels of cartilage-specific and inflammatory biomarkers, on the evaluation of pain and on the global patient assessment of disease activity.

This study demonstrated a statistically significant decrease of sColl2-1 cartilage specific biomarker, an early decrease of the ultrasensitive C-reactive protein (CRP), an improvement of the global assessment of the disease by the patient as well as a good tolerance and compliance for the treatment. Results of this exploratory study are encouraging and justify the setup of a randomized, placebo-controlled double blind and dose-ranging trial.

DETAILED DESCRIPTION:
150 patients suffering from symptomatic knee OA will be randomized in 3 parallel groups (50 patients per group). Each patient will be enrolled in the study for 6 months including 4 visits: Inclusion visit (T0), follow-up visits after 1 month (T1), 3 months (T3) and 6 months (T6).

A. Primary objective

- Evaluate the efficacy of two different dosages of FLEXOFYTOL® versus PLACEBO on arthritis related biomarker coll2-1 and on patient assessment of disease activity in patients suffering from knee OA after a 3 months treatment

B. Secondary objectives

* Evaluate the efficacy of two different dosages of FLEXOFYTOL® versus PLACEBO on arthritis-related and inflammatory biomarkers.
* Evaluate the efficacy of two different dosages of FL EXOFYTOL® versus PLACEBO on pain and function.
* Evaluate the tolerance, the compliance and the patients' satisfaction.
* Evaluate the use of rescue treatments i.e. Paracetamol and oral non-steroidal antiinflammatory drugs (NSAIDs) during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the age of 45 and 80

Exclusion Criteria:

* Artialis (study coordinator) or Tilman (Sponsor) 's employees
* Participation to a therapeutic clinical trial in the last 3 months
* Under guardianship or judicial protection

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-05; Primary Completion 2017-07 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Variation of serum levels of sColl2-1 biomarker between T0 and T3 by specific immunoassays (Enzyme-linked Immunosorbent assay, ELISA). | 3 months (between T0 and T3 visit)
Variation of Global assessment of disease activity by the patient using a Visual analogue scale (VAS) between T0 and T3. | 3 months (between T0 and T3 visit)

SECONDARY OUTCOMES:
Variation of serum levels of sColl2-1 (type II collagen degradation) and ultrasensitive CRP (C-reactive protein) biomarkers by specific immunoassays (Enzyme-linked Immunosorbent assay, ELISA). | 6 months (between T0 and T6 visit)
Mean knee pain over the last 24 hours using a visual analogue scale (VAS). | 6 months (between T0 and T6 visit)
Global assessment of disease activity using a visual analogue scale (VAS). | 6 months (between T0 and T6 visit)
Evaluation of Incidence of Emergent Adverse Events (AE), drop-outs and safety issues using blood safety analyses on patients with AE (Tolerance). | 6 months (between T0 and T6 visit)
Count the capsules in investigation kits brought back by the patient. | 6 months (between T0 and T6 visit)
Dosage by UHPLC-MS/MS and monitoring of curcumin blood level to assess patient compliance. | 6 months (between T0 and T6 visit)
Evaluation of Patient's satisfaction by Likert scale. | 6 months (between T0 and T6 visit)
Evaluate the use of rescue treatments i.e. Paracetamol and oral non-steroidal anti-inflammatory drugs (NSAIDs) during the study. | 6 months (between T0 and T6 visit)
Secondary outcome 8: Knee injury Osteoarthritis Outcome Score (KOOS) index and its subscale scores using a self-administered questionnaire. | 6 months (between T0 and T6 visit)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Liège (CHU-Liège)-Coordinating Center, Liège, Province of Liege, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henrotin Y, Malaise M, Wittoek R, de Vlam K, Brasseur JP, Luyten FP, Jiangang Q, Van den Berghe M, Uhoda R, Bentin J, De Vroey T, Erpicum L, Donneau AF, Dierckxsens Y. Bio-optimized Curcuma longa extract is efficient on knee osteoarthritis pain: a double-blind multicenter randomized placebo controlled three-arm study. Arthritis Res Ther. 2019 Jul 27;21(1):179. doi: 10.1186/s13075-019-1960-5. PMID 31351488
- See also: Decrease of a specific biomarker of collagen degradation in osteoarthritis, Coll2-1, by treatment with highly bioavailable curcumin during an exploratory clinical trial — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4032499/